CLINICAL TRIAL: NCT00871533
Title: Pilot Analysis of the Effects of IFN α2b Upon the Molecular Profile of Regional Lymph Nodes in Melanoma Patients With and Without Tumor-Involved Sentinel Lymph Nodes
Brief Title: Pilot Study of IFN α2b for Melanoma Patients
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Principal Investigator, Ahmad Tarhini, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-067
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Melanoma
Keywords: Biochemical Marker; Biochemical Markers; Biologic Marker; Biologic Markers; Biomarkers; Clinical Marker; Clinical Markers; Immune Marker; Immune Markers; Immunologic Marker; Immunologic Markers; Laboratory Marker; Laboratory Markers; Marker, Biochemical; Marker, Biological; Marker, Clinical; Marker, Immunologic; Marker, Laboratory; Marker, Serum; Marker, Surrogate; Markers, Biochemical; Markers, Biological; Markers, Clinical; Markers, Immunologic; Markers, Laboratory; Markers, Serum; Markers, Surrogate; Markers, Viral; Serum Marker; Serum Markers; Surrogate End Point; Surrogate End Points; Surrogate Endpoint; Surrogate Endpoints; Surrogate Marker; Surrogate Markers; Viral Marker; Viral Markers
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): REGIONAL PEG IFN MAINTENANCE: Regional PEG IFN-a2b given subcutaneously at "MAINTENANCE" dose level. (This arm has completed enrollment; non-evaluable subjects as defined in section 9.5 may be replaced at any point during study.
  Interventions: Drug: IFNα2b
- 2 (Experimental): No intervention / no injection control.
  Interventions: Drug: IFNα2b
- 3 (Experimental): PEG IFN INDUCTION: System PEG IFN-a2b given subcutaneously at "INDUCTION" dose level
  Interventions: Drug: PEG- IFNα2b
- 4 (Experimental): REGIONAL HDI MAINTENANCE: Regional HDI given subcutaneously at "MAINTENANCE" dose level per standard HDI regimen
  Interventions: Drug: PEG- IFNα2b
- 5 (No Intervention): HDI Induction: Systemic HDI given intravenously at "INDUCTION" dose level per the standard HDI regimen.

INTERVENTIONS:
Drug: IFNα2b — IV injection at 20 million IU/m2. IFNα2b IV injection will be performed every day between day -14 and day -9 (5 infusions) and also every day between day -7 and day -2 (5 infusions) for a total of 10 infusions.
  Arms: 1
Drug: IFNα2b — SC injections peri-lesionally (PL) in the vicinity of the primary, at 10 million IU/m2. IFNα2b Injection will be performed every other day between day -14 and day -9 (3 injections) and also every other day between day -7 and day -2 (3 injections) for a total of 6 injections.
  Arms: 2
Drug: PEG- IFNα2b — SC injection at 6mcg/kg will be performed systemically (at site that is not regional): first injection at day -14, second injection at day -7, for a total of 2 injections.
  Arms: 3
Drug: PEG- IFNα2b — SC injections peri-lesionally (PL) in the vicinity of the primary at 3ug/kg: first injection at day -14, second injection at day -7, for a total of 2 injections.
  Arms: 4

SUMMARY:
The presence of malignant cells in lymph nodes is a critical parameter in the staging of melanoma cancer patients. Assessment of lymph nodes is currently done by histopathology alone. The long-term survival of melanoma cancer patients who have Stage IB disease (no known lymph node involvement with a tumor greater than 2 cm) is lower than patients who are Stage IA (no known lymph node involvement with a tumor less than 2 cm). Likewise, the survival rates of patients who are judged to be Stage II based on histologically positive level-one lymph nodes is often no better than that of higher stage patients who have level-two lymph node involvement. These observations suggest that micrometastases are often present in lymph nodes that are not detectable by histological assessment.

The collection of Sentinel Lymph Nodes (SLN) and non SLN material outlined in this proposal will permit both targeted and exploratory studies, without compromising the patient's diagnosis, on specimens that represent central engines of the immune response and whose function in the context of tumor progression is largely unknown.

With the advent of an array of new methodologies that utilize minimum material for both molecular and cellular assessments, acquiring up to 20% and in general the investigators anticipate the use of 5% on average of SLN and/or non SLN tissue for research purposes, may prove to be critical to understanding the impact of nodal tumor involvement on patient outcome and survival.

ELIGIBILITY:
Inclusion Criteria:

* Primary melanoma with the following Breslow thickness and stage

  * less than or equal to 2 mm
  * Patients with recent (within 12 wks) biopsy of primary melanoma that has not been widely resected will be eligible for study according to the above-specified criteria for tumor thickness and stage.
* Age 18 years or older.
* Patients must have documented hemoglobin level of 10g/dL or higher and normal organ function tests including BUN, Creatinine, and liver enzyme panel to include AST, ALT, and Bilirubin. This can be drawn on the day of consent, or be documented from a previous visit within the past 30 days
* Negative serum pregnancy test
* Subjects must have provided written, informed consent prior to any study procedures: collection of blood and LN tissue specimens for this protocol.

Exclusion Criteria:

* Serious illnesses, such as: cardiovascular disease (uncontrolled congestive heart failure, hypertension, cardiac ischemia, myocardial infarction, severe cardiac arrhythmia), bleeding disorders, autoimmune diseases, severe obstructive or restrictive pulmonary diseases, active systemic infections, inflammatory bowel disorders, severe renal disease.
* Any significant psychiatric disease, medical intervention, or other condition, which in the opinion of the Principal Investigator or Co-Investigators, could prevent adequate informed consent or compromise participation in the clinical trial.
* Active infection or antibiotics within one-week prior to study.
* Systemic steroid or other immunosuppressive therapy administered for more than 10 days within 4 weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
To utilize gene-profiling analysis of regional lymph node tissue to molecularly characterize the effect of IFN α2b and PEG IFNα2b on the SLN. Endpoint: mRNA expression by gene array. | 5

SECONDARY OUTCOMES:
Quantitate putative biomarkers differentially expressed in the SLN for each active treatment group and among all active treatment groups combined. Endpoint: mRNA expression by Taqman. | 5
Molecularly characterize the effect of perilesional IFN α2b and PEG IFNα2b administered as close as possible to the primary tumor site on SLNs that are positive vs. negative for tumor micrometastases. Endpoint: mRNA expression by gene array. | 5

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States